CLINICAL TRIAL: NCT02496611
Title: Enhancing Weight Loss Maintenance With GLP-1RA (BYDUREON™) in Adolescents With Severe Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1505M72081
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Severe Obesity
Keywords: Obesity; Pharmacotherapy; GLP-1; Children; Exenatide; BYDUREON; Weight Loss; Maintenance
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Individuals who consented to the project were enrolled in a screening phase of the study where they received meal replacement therapy in attempt to achieve a >/= 5% body mass reduction. Individuals who did not meet this goal were considered screen failures. Individuals who met this goal were allowed to remain in the study and be randomized to one of the treatment arms (placebo or GLP-1 RA).
  A total of 100 participants consented and were enrolled and 66 participants achieved the required BMI reduction with MRT and were randomized to study treatment (33 to GLP-1 RA (exenatide) and 33 to placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight Loss Maintenance without Pharmacotherapy (Placebo Comparator): Individuals who, after a short-term (1-3 month) meal replacement induction period, achieve ≥5% BMI reduction. A selection of these participants are then randomized to receive treatment with placebo.
  Interventions: Drug: Weight loss without pharmacotherapy
- Weight Loss Maintenance with Pharmacotherapy (Active Comparator): Individuals who, after a short-term (1-3 month) meal replacement induction period, achieve a >/= 5% BMI reduction. A selection of these participants are then randomized to receive treatment with GLP-1RA.
  Interventions: Drug: Weight loss with pharmacotherapy

INTERVENTIONS:
Drug: Weight loss with pharmacotherapy — Participants randomized to the drug intervention group will receive Exenatide extended-release.
  Other Names: Exenatide extended release
  Arms: Weight Loss Maintenance with Pharmacotherapy
Drug: Weight loss without pharmacotherapy — Participants randomized to the placebo group will receive a placebo.
  Other Names: Placebo
  Arms: Weight Loss Maintenance without Pharmacotherapy

SUMMARY:
Long-term weight loss maintenance is seldom achieved by individuals with obesity owing to numerous biological adaptations involving appetite, satiety, and energy expenditure in the post- weight loss setting. Following a loss in body weight, peripheral and central mechanisms convey a sense that energy reserves have dwindled, activating a strong counter response to increase caloric intake. Adolescents with severe obesity are not immune to the vexing issue of weight regain. Indeed, only 2% are able to achieve and maintain clinically-meaningful weight loss with lifestyle modification therapy. Therefore, novel treatment paradigms focused on long-term weight loss maintenance are urgently needed. Pharmacotherapy has the potential to prevent weight regain by targeting specific counter-regulatory mechanisms in the post- weight loss setting. One of the most promising candidates is the glucagon like peptide-1 receptor agonist (GLP-1RA) class, which greatly enhanced weight loss maintenance following a short-term low calorie diet among adults with obesity. The rationale for focusing on GLP-1RA treatment (BYDUREON™) to prevent weight regain is supported by the multiple central and peripheral mechanisms of action targeted by this class of drug; many of which specifically address the biological adaptations known to induce relapse. The investigators have strong preliminary data demonstrating that GLP-1RA treatment reduces BMI in adolescents with severe obesity. Moreover, the investigators and others have shown that although meal replacement therapy (structured meals of known caloric content) can elicit robust short-term weight loss among adolescents with severe obesity, weight regain is a pervasive problem. Therefore, in this clinical trial, our innovative approach will utilize GLP-1RA treatment to target weight regain following short-term meal replacement therapy in youth with severe obesity. Participants who achieve ≥5% BMI reduction during the meal replacement phase will be randomized to GLP-1RA treatment or placebo for an additional 52 weeks while simultaneously engaging in lifestyle modification therapy. Importantly, this study will also allow us to examine the extent to which GLP-1RA treatment addresses mechanisms of weight regain, investigate other pleiotropic benefits of GLP-1RA, and identify predictors of weight loss response.

DETAILED DESCRIPTION:
Primary Objective Evaluate the effect of GLP-1RA treatment on the maintenance of weight loss and durability of cardiometabolic risk factor improvements among adolescents with severe obesity following a meal replacement induction period. The investigators hypothesize that adolescents with severe obesity receiving GLP-1RA treatment following a short-term meal replacement induction period will demonstrate superior maintenance of initial BMI reduction 52 weeks following randomization compared to those assigned to placebo (primary endpoint) and that a higher proportion of those assigned to GLP-1RA treatment vs. placebo will maintain ≥5% BMI reduction from baseline to the 52-week time point (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥1.2 times the 95th percentile (based on sex and age) or BMI ≥35 kg/m2
* 12-17 years old

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Previous (within 6 months) or current use of medication(s) prescribed primarily for weight loss (refer to appendix material for comprehensive list)
* If currently using weight altering drug(s) for non-obesity indication(s) (refer to appendix material for comprehensive list), any change in drug(s) or dose within the previous 6 months
* Previous bariatric surgery
* If currently using anti-hypertensive medication(s), lipid medication(s), and/or medication(s) to treat insulin resistance (refer to appendix material for comprehensive list), any change in drug(s) or dose within the previous 6 months
* If currently using CPAP/BIPAP (for sleep apnea), change in frequency of use or settings within the previous 6 months
* History of treatment with growth hormone
* Neurodevelopmental disorder severe enough to impair ability to comply with study protocol
* Clinical diagnosis of bipolar illness, schizophrenia, conduct disorder, and/or substance use/abuse
* Females: currently pregnant, planning to become pregnant, or unwilling to use 2 or more acceptable methods of contraception when engaging in sexual activity throughout the study
* Tobacco use
* Liver/renal dysfunction
* ALT or AST >2 times the upper limit of normal
* Bicarbonate <18 mmol/L
* Creatinine >1.2 mg/dL
* History of pancreatitis
* Personal- and/or family history of medullary thyroid carcinoma
* Personal- and/or family history of multiple endocrine neoplasia type 2
* Calcitonin level >50 ng/L
* Bulimia nervosa
* Neurological disorder
* Hypothalamic obesity
* Obesity associated with genetic disorder (monogenetic obesity)
* Hyperthyroidism or uncontrolled hypothyroidism
* History of suicide attempt
* History of suicidal ideation or self-harm within the past year
* History of cholelithiasis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Fox CK, Clark JM, Rudser KD, Ryder JR, Gross AC, Nathan BM, Sunni M, Dengel DR, Billington CJ, Bensignor MO, Kelly AS. Exenatide for weight-loss maintenance in adolescents with severe obesity: A randomized, placebo-controlled trial. Obesity (Silver Spring). 2022 May;30(5):1105-1115. doi: 10.1002/oby.23395. Epub 2022 Apr 10. PMID 35403350
- [Derived] Ryder JR, Kaizer AM, Rudser KD, Daniels SR, Kelly AS. Utility of Body Mass Index in Identifying Excess Adiposity in Youth Across the Obesity Spectrum. J Pediatr. 2016 Oct;177:255-261.e2. doi: 10.1016/j.jpeds.2016.06.059. Epub 2016 Aug 2. PMID 27496270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 participants consented to enroll in the study and entered the screening phase. During the screening phase participants entered and 8-week meal replacement therapy phase to help them meet a goal of achieving reducing their body mass by 5% or more. Only those participants who met this weight loss goal passed the study screening and were allowed to be randomized to receive placebo or GLP-1 RA. 66 participants met the BMI weight loss goal, 34 participants did not pass the screening phase.
Pre-assignment Details: Only individuals who achieve the >/= 5% BMI reduction will be considered to have passed screening and will be allowed to be randomized to treatment with GLP-1 RA or placebo.
Groups:
- Weight Loss Maintenance Without Pharmacotherapy: A total of 33 participants who met the initial weight loss goal during the meal replacement induction were randomized to receive lifestyle therapy and placebo.
- Weight Loss Maintenance With Pharmacotherapy: A total of 33 participants who met the initial weight loss goal during the meal replacement induction were randomized to receive lifestyle therapy and pharmacotherapy with Exenatide extended-release.
Period: Overall Study
Arm/Group | Weight Loss Maintenance Without Pharmacotherapy | Weight Loss Maintenance With Pharmacotherapy
Started | 33 | 33
Completed | 26 | 30
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Weight Loss Maintenance Without Pharmacotherapy: A short-term (1-3 month) meal replacement induction period design to achieve ≥5% BMI reduction. If participants achieve ≥5% BMI they will be randomized to drug or placebo in phase 2 of the trail.
  Meal Replacement Therapy: A short-term meal replacement induction period designed to achieve >5% BMI reduction in 1, 2, or 3 months.
- Weight Loss Maintenance With Pharmacotherapy: We hypothesize that adolescents with severe obesity receiving GLP-1RA treatment following a short-term meal replacement induction period will demonstrate superior maintenance of initial BMI reduction 52 weeks following randomization compared to those assigned to placebo (primary endpoint) and that a higher proportion of those assigned to GLP-1RA treatment vs. placebo will maintain ≥5% BMI reduction from baseline to the 52-week time point (secondary endpoint)
  Exenatide extended-release for injectable suspension (BYDUREON™)
- Total: Total of all reporting groups
Arm/Group | Weight Loss Maintenance Without Pharmacotherapy | Weight Loss Maintenance With Pharmacotherapy | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 33 | 66
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 20 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 31 | 27 | 58
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index
Description: Percentage of body mass index change from Randomization to Week 52
Time Frame: 52 weeks
Population: Change in body mass index (percentage) from Randomization to Week 52.
Measure: Mean (Standard Deviation); unit: percentage (body mass index)
Groups:
- Weight Loss Maintenance Without Pharmacotherapy: A short-term (1-3 month) meal replacement induction period design to achieve ≥5% BMI reduction. If participants achieve ≥5% BMI they will be randomized to drug or placebo in phase 2 of the trial.
  Individuals in this group were randomized to receive lifestyle management therapy with placebo.
- Weight Loss Maintenance With Pharmacotherapy: A short-term (1-3 month) meal replacement induction period design to achieve ≥5% BMI reduction. If participants achieve ≥5% BMI they will be randomized to drug or placebo in phase 2 of the trial.
  Individuals in this group were randomized to receive lifestyle management therapy with pharmacotherapy treatment with Exenatide extended-release.
Arm/Group | Weight Loss Maintenance Without Pharmacotherapy | Weight Loss Maintenance With Pharmacotherapy
Number analyzed (Participants) | 33 | 33
percentage (body mass index) | 10.1 (9.0) | 4.6 (10.5)

ADVERSE EVENTS:
Time Frame: Adverse event and serious adverse event data was collected from Baseline to Week 52.
Description: The adverse events and serious adverse events that are reported are for those participants who met the minimum 5% BMI loss goal and were eligible to be randomized to receive either the placebo or GLP-1 RA.
Groups:
- Weight Loss Maintenance Without Pharmacotherapy: A short-term (1-3 month) meal replacement induction period design to achieve ≥5% BMI reduction. If participants achieve ≥5% BMI they will be randomized to drug or placebo in phase 2 of the trial.
  Individuals in this group were randomized to receive lifestyle maintenance therapy without pharmacotherapy.
  Serious Adverse Events and Adverse Events were not reported during the meal replacement induction.
- Weight Loss Maintenance With Pharmacotherapy: A short-term (1-3 month) meal replacement induction period design to achieve ≥5% BMI reduction. If participants achieve ≥5% BMI they will be randomized to drug or placebo in phase 2 of the trial.
  Individuals in this group were randomized to receive lifestyle maintenance therapy with pharmacotherapy.
  Serious Adverse Events and Adverse Events were not reported during the meal replacement induction.
- Meal Replacement Induction: A short-term (1-3 month) meal replacement induction period to achieve ≥5% BMI reduction. If participants achieve ≥5% BMI they will be randomized to drug or placebo in phase 2 of the trial.
  All individuals were enrolled into this group upon signing consent and determining eligibility.
  Serious Adverse Events and Adverse Events were not reported during the meal replacement induction.
Arm/Group | Weight Loss Maintenance Without Pharmacotherapy | Weight Loss Maintenance With Pharmacotherapy | Meal Replacement Induction
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/33 | 0/100
Other Adverse Events (participants affected / at risk) | 30/33 | 32/33 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss Maintenance Without Pharmacotherapy (N=33) | Weight Loss Maintenance With Pharmacotherapy (N=33) | Meal Replacement Induction (N=100)
Hospitalization for chemical dependency (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA — One participant who had been randomized to Exenatide extended-release was hospitalized for chemical dependency treatment after a drug (not related to the study) and alcohol overdose.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss Maintenance Without Pharmacotherapy (N=33) | Weight Loss Maintenance With Pharmacotherapy (N=33) | Meal Replacement Induction (N=100)
Nausea (Gastrointestinal disorders) | 7 (7) | 13 (15) | NA
Vomiting (General disorders) | 2 (3) | 13 (15) | NA
Diarrhea (Hepatobiliary disorders) | 6 (6) | 11 (14) | NA
Constipation (Hepatobiliary disorders) | 6 (9) | 6 (6) | NA
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 5 (5) | NA
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (4) | NA
Dizziness (Nervous system disorders) | 3 (3) | 4 (4) | NA
Flu-like symptoms (Immune system disorders) | 4 (4) | 3 (3) | NA
Headache (General disorders) | 14 (17) | 19 (20) | NA
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 24 (29) | 26 (32) | NA
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 7 (7) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT02496611/Prot_SAP_000.pdf